CLINICAL TRIAL: NCT00121186
Title: Nonmyeloablative Allogeneic Stem Cell Transplantation For Relapsed Hodgkin's or Non-Hodgkin's Lymphoma After Autologous Transplantation ( A BMT Study)
Brief Title: S0501 Fludarabine, Melphalan, and Donor Stem Cell Transplant Followed By Tacrolimus and Methotrexate in Treating Patients for Relapsed Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000435930; S0501 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent small lymphocytic lymphoma; recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — fludarabine phosphate; Melphalan; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nonmyeloablative allogeneic stem cell transplant (Experimental): Patients are given fludarabine 30 mg/m^2 on days -6 to -2 and melphalan 70 mg/m^2 on days -3 and -2, then transplanted with donor peripheral blood stem cells or harvested bone marrow stem cells on day 0. Patients are then given post-transplant immunosuppression consisting of tacrolimus 0.06 mg/kg/day on days -3 to 100 and methotrexate 5 mg/m^2 on days 1, 3, and 7.
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Drug: methotrexate; Drug: tacrolimus; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: fludarabine phosphate — 30 mg/m^2 on days -6 to -2 (2-6 days before transplant).
Drug: melphalan — 70 mg/m^2 on days -3 and -2 (2-3 days before transplant).
Drug: methotrexate — 5 mg/m^2 on days 1, 3, and 7 post-transplant.
Drug: tacrolimus — 0.03 mg/kg bid on days -3 to 100 post-transplant.
Procedure: allogeneic bone marrow transplantation — if donor bone marrow stem cells are harvested
Procedure: peripheral blood stem cell transplantation — if donor peripheral blood stem cells are harvested

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and melphalan, before a donor bone marrow or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and methotrexate after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine together with melphalan followed by tacrolimus and methotrexate works in treating patients who are undergoing a donor stem cell transplant for relapsed lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 1-year progression-free and overall survival rate in patients with relapsed Hodgkin's or non-Hodgkin's lymphoma after prior autologous stem cell transplantation treated with a nonmyeloablative conditioning regimen comprising fludarabine and melphalan followed by allogeneic bone marrow or peripheral blood stem cell transplantation and immunosuppression comprising tacrolimus and methotrexate.
* Determine treatment-related mortality in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine engraftment of donor hematopoietic stem cells, as measured by hematopoietic recovery and donor-derived hematopoiesis (determined by T cell and neutrophil specific chimerism) at 2, 3, 6, and 12 months, in patients treated with this regimen.
* Determine the incidence of acute and chronic graft-versus-host disease in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (Hodgkin's lymphoma vs non-Hodgkin's lymphoma).

Patients receive fludarabine IV over 1 hour on days -6 to -2 and melphalan IV over 15-20 minutes on days -3 and -2. Patients undergo allogeneic peripheral blood stem cell or bone marrow transplantation on day 0. Patients receive oral tacrolimus twice daily beginning on day -3 and continuing until day 100 followed by a taper to day 180. Patients also receive methotrexate IV on days 1, 3, and 7. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study transplantation, patients are followed at 1 and 3 months, 1 year, and then annually for up to 4 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of lymphoma of 1 of the following types:

  * Diffuse large B-cell lymphoma
  * Follicular lymphoma

    * Grades 1, 2, or 3
  * Primary mediastinal lymphoma
  * Mantle cell lymphoma
  * Small lymphocytic lymphoma
  * Hodgkin's lymphoma
  * Transformed lymphoma
* Relapsed after prior autologous bone marrow transplantation (BMT)

  * More than 180 days post BMT
* Received ≥ 1 course of chemotherapy after BMT relapse

  * Achieved a complete response OR a partial response to chemotherapy

    * Largest residual tumor dimension ≤ 2 cm
* No clinical or laboratory evidence of CNS involvement by lymphoma
* HLA-identical donor available, meeting 1 of the following criteria:

  * Sibling donor with 5/6 or 6/6 alleles matching by genotyping

    * No monozygotic identical twins
  * Unrelated donor with 10/10 alleles matching by genotyping

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* LVEF ≥ 40% by MUGA or 2-D echocardiogram (2-D ECHO)
* No significant cardiac abnormalities by MUGA or 2-D ECHO
* No uncompensated coronary artery disease by ECG or physical exam
* None of the following within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Uncontrolled atrial fibrillation
* None of the following within the past 3 months:

  * Severe peripheral vascular disease
  * Venous stasis ulcers
  * Deep venous or arterial thrombosis
* No uncontrolled hypertension

Pulmonary

* DLCO (corrected) and total lung capacity ≥ 40% of predicted
* No requirement for continuous supplemental oxygen

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No AIDS
* No active bacterial, viral, or fungal infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of uncontrolled seizures
* No diabetic ulcers within the past 3 months

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No more than 1 prior bone marrow transplantation

Chemotherapy

* See Disease Characteristics
* More than 21 days since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior major surgery except placement of a venous access device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Stiff, MD, Study Chair — Loyola University; Scott E. Smith, MD, PhD, FACP, Study Chair — Loyola University
Locations (33):
- United States (33):
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nonmyeloablative Allogeneic Stem Cell Transplant
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nonmyeloablative Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 1
Age Continuous [Median (Full Range); unit: years] | 47.2 [47.2 to 47.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS rate at 1 year.
Time Frame: 1, 3, and 12 months after protocol treatment, then every 3 months for 1 year, every 6 months for year 2, then annually thereafter until 5 years after registration
Measure: Number; unit: participants
Arm/Group | Nonmyeloablative Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 1
participants | 1

2. Primary Outcome: Overall Survival
Description: OS rate at 1 year.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nonmyeloablative Allogeneic Stem Cell Transplant
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: After transplant, and after every month of protocol treatment, for a maximum of 6 months
Arm/Group | Nonmyeloablative Allogeneic Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nonmyeloablative Allogeneic Stem Cell Transplant (N=1)
Hemoglobin (Blood and lymphatic system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Platelets (Investigations) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No